CLINICAL TRIAL: NCT03106207
Title: Prospective Single-center Study to Evaluate Preoperative and Postoperative Endoscopic Alterations in Patients Submitted to Gastric Bypass Without a Ring.
Brief Title: Preoperative and Postoperative Endoscopic Alterations in Patients Submitted to Gastric Bypass Without a Ring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KaiserCDH
Record Dates: First submitted 2017-03-12; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper gastric endoscopy (UGE) (Other): Patients will be submitted to a UGE before the gastric bypass surgery without a ring and at two, six and 12 months after the surgical procedure .
  Interventions: Procedure: Upper gastric endoscopy (UGE)

INTERVENTIONS:
Procedure: Upper gastric endoscopy (UGE) — UGE will be performed before the gastric bypass surgery and post-surgery at two, six and 12 months of clinical visit.

SUMMARY:
Despite the high success rates of gastric bypass in the short and long terms, little is known about possible anatomopathological changes that can occur in these patients. The objective is to investigate preoperative and postoperative endoscopic changes in patients undergoing gastric bypass without a ring. Thirty obese patients from different regions of the country with the surgical indication for the Roux-en-Y gastric bypass will be studied prospectively. All patients will be submitted to upper gastric endoscopy (UGE) two, six and 12 months after the surgical procedure at the Kaiser Clinic. This study will identify whether there are endoscopic changes within one year after the surgery and what they are. Changes, if they exist, will be correlated with clinical data, in order to make an accurate prognosis of the patient, thereby contributing to the outcomes of future patients submitted to this type of procedure.

DETAILED DESCRIPTION:
People with severe or morbid obesity often fail to lose weight in the long term. Gastric bypass is considered the gold standard in the surgical treatment of obesity. Despite the high success rates of gastric bypass in the short and long terms, little is known about possible anatomopathological changes that can occur in these patients. UGE has been used on a wide scale in complementary evaluations of patients submitted to bariatric surgery. However, there is still no consensus on the use of imaging tests such as UGE in the follow-up of these patients after surgery. Considering the importance of gastric bypass in the treatment of obesity, knowledge about possible preoperative and postoperative GI alterations identified by endoscopy in these patients may contribute to the establishment of correlations with symptomatology and with the success rate of this technique during follow-ups of up to 12 months.

Organization and infrastructure: This study is organized based on a single location: the Kaiser Clinic and Day Hospital. This center is renowned for the treatment of diseases in the areas of Gastroenterology, Proctology and General Surgery.

Objectives:

General: Demographic, clinical, nutritional, operative and endoscopic data will be assessed.

Specific: The objective of this research will be to investigate preoperative and postoperative endoscopic changes in patients undergoing gastric bypass without a ring.

Patients and Methods: Thirty obese patients from different regions of the country with surgical indication for the Roux-en-Y gastric bypass will be studied prospectively. Patients who meet the inclusion criteria will be invited to participate and, on agreeing, they will sign Informed Consent Forms. The procedures will be performed only after patients give their written consent.

Clinical evaluation of the patients Clinical history: Patients will be questioned about the frequency and intensity of their symptoms. Commonly used medications will be noted as well as drugs used for symptomatic relief (number of tablets). Any urgent/emergency events (such as emergency room visits and/or hospital admission) will be investigated. Other clinical events will also be recorded.

Physical examination:A physical examination (general and gastroenterological) will be performed routinely in all patients participating in this study.

Procedures in the pre- and post-procedure phases: Patients will be submitted to a UGE before the gastric bypass surgery without a ring. All changes related to the esophageal body, distal esophagus and stomach will be analyzed. Biopsies will be performed of the distal esophagus (two fragments 4 cm above the esophagogastric transition), gastric body (anterior and posterior walls), incisura angularis and gastric antrum (large and small pre-pyloric curvature). Furthermore, biopsies will be performed of any lesions detected in the esophagus or stomach.

All patients will be submitted to UGE two, six and 12 months after the surgical procedure. The following will be performed in postoperative endoscopies:

1- The mucosa of the esophageal body will be studied, biopsies of the distal esophagus (two fragments) and small curvature (two fragments) will be performed and the gastric pouch width and anteroposterior diameter and length of the small curvature will be evaluated; 2 - the shape of the gastrojejunal anastomosis will be evaluated and the maximum diameter will be measured and 3 - the jejunal loops will be studied in relation to mucosal changes and afferent loop size and angulation.

All exams will be performed at the Kaiser Clinic after patients have fasted for at least eight hours and signed an informed consent form for the UGE. With the patient in left lateral decubitus position, 10% xylocaine spray will be instilled followed by 50 mcg fentanyl EV and 5 mg midazolam EV. After sedation, an Olympus CV 180 endoscope (Olympus, Tokyo, Japan) will be introduced orally. The images obtained will be transferred to a Olympus EVIS EXERA II processor connected to a computer unit with the ZScan 5 program (Zscan Software Ltda, Goiânia, Brazil). When the patient regains his level of consciousness, he will be released in the company of a responsible adult.

Postoperative clinical evaluation: After hospital discharge, all patients should return for outpatient follow-ups including a clinical evaluation and endoscopy exams.

Clinical visits will be scheduled as follows:

Visit 1 - 2 months; Visit 2 - 6 months; Visit 3 - 12 months

Clinical complications / adverse events / clinical outcomes: For all patients, any possible clinical complication will be promptly checked by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and younger than 65 years of age;
* Patients with indication for gastric bypass without ring;
* Patient attending regular appointments in the Gastroenterology Service.

Exclusion Criteria:

* Patients younger than 18 and over 65 years of age;
* Patients who have no indication of gastric bypass without a ring;
* Pregnant women (a BHCG test will be required from all women of childbearing age).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2016-12-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | Before surgery and at 2, 6, 12 and 24 months
  weight in kg

SECONDARY OUTCOMES:
The mucosal lesions of the distal esophageal body by Los Angeles Classification | Before surgery and at 2, 6, 12 and 24 months
  The biopsies of the distal esophagus (two fragments) will be performed to study the mucosa through upper gastric endoscopy.
Gastric pouch Anteroposterior diameter (cm) | Before surgery and at 2, 6, 12 and 24 months
  All measurements will be evaluated through UGE
Length of lesser curvature (cm) | Before surgery and at 2, 6, 12 and 24 months
  All measurements will be evaluated through UGE
Gastrojejunal anastomosis (mm) | Before surgery and at 2, 6, 12 and 24 months
  All measurements will be evaluated through UGE
The mucosal changes in jejunal loops will be studied for any lesion like marginal ulcers | Before surgery and at 2, 6, 12 and 24 months
  The mucosal changes will be evaluated through UGE
Quality of Afferent loop size as adequate or not. | Before surgery and at 2, 6, 12 and 24 months
  Afferent loop size will be evaluated through UGE
Afferent loop angulation | Before surgery and at 2, 6, 12 and 24 months
  Evaluated through UGE: the Y (two bowel) afferent bowel or efferent bowel

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Gustavo de Quadros, MD, Principal Investigator — Kaiser Clinica and Day Hospital
Locations (1):
- Kaiser Clinic and Day Hospital, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided